CLINICAL TRIAL: NCT02586532
Title: Evaluation of the Sensitivity of Endoscopy to Detect Nasopharyngeal Carcinoma (NPC) in an Epstein-Barrr Virus (EBV)-Based NPC Screening Project in China
Brief Title: Evaluation of the Sensitivity of Endoscopy to Detect Nasopharyngeal Carcinoma (NPC) in an Epstein-Barr Virus (EBV)-Based NPC Screening Project in China
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916007; 16-C-N007
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: Detection; Cancer; Antibody; Biopsy; Registry
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Residents of towns participating in China Demonstration Project.

SUMMARY:
Background:

Epstein-Barr virus (EBV) can cause the cancer nasopharyngeal carcinoma (NPC). Early detection of NPC through screening can lead to better treatment outcomes than when it is found later. Currently, NPC is found through visual inspection with an endoscope. It is not clear how well this method works, especially for the identification of small, early cancers. Researchers want to see how well nasal endoscopy works to detect NPC compared to another method called magnetic resonance imaging (MRI).

Objectives:

To evaluate the sensitivity of endoscopy to detect prevalent NPC among people who screen positive for EBV antibodies.

Eligibility:

Participants of the NPC Early Detection Screening Program in China who:

Have increased levels of EBV antibodies

Are otherwise in good health and able to have an MRI procedure

Design:

Participants will be screened with a blood test.

Participants will have a nasal endoscopy.

Participants will have an MRI of the head and neck:

Participants will have lesions identified by either the endoscopy or MRI biopsied and sent to a pathologist for review and diagnosis of NPC.

Researchers will compare NPC detection rates by endoscopy and by MRI to see which method is better able to identify prevalent NPC.

...

DETAILED DESCRIPTION:
Epstein-Barr virus (EBV) is a necessary cause of nasopharyngeal carcinoma (NPC). Individuals who develop NPC have been shown to have an altered EBV antibody profile. Ongoing efforts to evaluate EBV antibody testing as a screening test for the early detection of NPC have been launched in China and Taiwan but it is unclear whether the current method to detect NPC among screen-positive individuals (i.e., visual inspection with the aide of an endoscope) is sufficiently sensitive to detect prevalent cancers among screen positive individuals. In the present study, we aim to evaluate the sensitivity of endoscopy to detect NPC. The study is embedded within a large, community-based trial in China to evaluate EBV antibody testing as a screening test that triages individuals into endoscopy for the early detection of NPC. We plan to enroll 1,000 individuals with elevated EBV antibody scores within the active screening arm of the trial in China. Participants will have both endoscopy and MRI performed to detect nasopharyngeal lesions. Lesions identified by either method will be biopsied and evaluated for the presence of NPC. NPC cases will also be identified by linkage to the regional cancer registry. We expect to identify a total of 25 histologically confirmed NPC cases through endoscopy, MRI and/or registry linkage. The sensitivity of endoscopy to detect prevalent NPC will be estimated. Characteristics of prevalent NPC cases detected by MRI or registry linkage but missed by endoscopy will be described, with respect to clinical stage, socio-demographic and other characteristics. This study is an important complement to the ongoing screening trial in China, as a highly sensitive EBV-based screening test can ultimately be successful only if methods available to identify cancer among screen-positive individuals are equally sensitive. Demonstration of high sensitivity of endoscopy to detect NPC will be reassuring. Demonstration of reduced sensitivity will trigger the need to consider alternatives to endoscopy for the diagnosis of NPC.

ELIGIBILITY:
* INCLUSION CRITERIA:

Already participating in the NPC Early Detection Screening Program;

Increased levels of EBV antibodies and referred for nasal endoscopy;

No metallic materials in the body;

Have a health examination score of 0 or 1;

Normal creatinine blood levels; and

For women, not pregnant.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of towns participating in China Demonstration Project.
Sampling Method: Probability Sample
Enrollment: 828 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Concordance of Endoscopy and MRI screening for NPC | ongoing
  NPC

CONTACTS AND LOCATIONS:
Overall Officials: Allan Hildesheim, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Sun Yat-sen University Cancer Center (SYSUCC), Guangzhou, China